CLINICAL TRIAL: NCT05283395
Title: A Multicenter, Open-Label Rocklatan® (Netarsudil/Latanoprost Ophthalmic Solution) 0.02%/0.005% Evaluation of IOP Lowering Efficacy and Safety as Replacement of Current Medical Therapy Regimen for the Reduction of Elevated Intraocular Pressure in Patients With Glaucoma or Ocular Hypertension
Brief Title: Rocklatan® Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-ROC-22-003
Record Dates: First submitted 2022-03-07; First posted 2022-03-17 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — netarsudil; Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rocklatan (Experimental): Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution, one drop in each eye in the evening for 12 weeks
  Interventions: Drug: Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution

INTERVENTIONS:
Drug: Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution — Commercially available ophthalmic solution indicated for the reduction of elevated intraocular pressure (IOP) in patients with open-angle glaucoma or ocular hypertension
  Other Names: Rocklatan®

SUMMARY:
The objective of this study is to evaluate the IOP-lowering effect when subjects are switched from various latanoprost-based regimens to Rocklatan. Subjects will stop their IOP-lowering medical therapy regimen and dose with Rocklatan for the duration of the study (12 weeks).

DETAILED DESCRIPTION:
Enrollment will be stratified according to subject's IOP-lowering medical therapy regimen as follows:

* Latanoprost monotherapy (Latanoprost Mono)
* Latanoprost plus 1 additional IOP-lowering agent (Latanoprost +1)
* Latanoprost plus 2 additional IOP-lowering agents (Latanoprost +2)

Aerie Pharmaceuticals was acquired by Alcon Research LLC on November 22, 2022.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects age 18 or older
* Current diagnosis of open-angle glaucoma or ocular hypertension
* Subject currently being treated with latanoprost alone or latanoprost plus 1 or 2 additional agents/bottles. Current IOP lowering regimen is stable for at least 30 days prior to Baseline Visit
* Treated IOP ≥ 20 mmHg measured in the morning (before noon) at the Baseline Visit by Goldmann applanation tonometer
* Best corrected Snellen visual acuity of 20/100 or better in both eyes
* Willingness to follow protocol requirements, including signed informed consent and health information release forms, routine follow-up schedule, completing questionnaires

Key Exclusion Criteria:

* Have any active ocular disease other than open-angle glaucoma or ocular hypertension that would interfere with study interpretation
* Use of fixed dose combination agents as part of the patient's Baseline IOP lowering therapy regimen, if not also on latanoprost
* Active ocular infection/inflammation or history of uveitis
* Aphakic or pseudophakic patients with a torn posterior lens capsule, or with known risk factors for macular edema
* Any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results
* Use of topical, periorbital, intravitreal or systemic steroid within previous 3 months or expected use during the course of the study
* Prior participation in any investigational drug or device study within the last 30 days prior to the Baseline Visit.
* Known sensitivity or allergy to the study medication or components
* Females who are pregnant, nursing, or planning a pregnancy during the study
* Positive pregnancy test at Baseline Visit (women of childbearing potential only)
* Women of childbearing potential who are not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Advisor, Clinical R&D, Study Director — Alcon Research, LLC
Locations (21):
- United States (21):
  - North Valley Eye Medical Group, Mission Hills, California
  - Visionary Eye Institute, Newport Beach, California
  - California Eye Specialists Medical Group, Pasadena, California
  - North Bay Eye Associates, Petaluma, California
  - Shettle Eye Research, Largo, Florida
  - Center For Sight, Venice, Florida
  - Georgia Eye Partners, Atlanta, Georgia
  - Coastal Research Associates LLC, Roswell, Georgia
  - Tekwani Vision Center, St Louis, Missouri
  - OCLI Vision, Manhasset, New York
  - Mark J. Weiss, MD, Inc., Tulsa, Oklahoma
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Advancing Vision Research, Goodlettsville, Tennessee
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Keystone Research, Austin, Texas
  - Louis M. Alpern, M.D., M.P.H., P.A, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Vistar Eye Center, Roanoke, Virginia
  - The Eye Centers of Racine and Kenosha, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 21 investigative sites located in the United States.
Pre-assignment Details: This reporting population includes all participants who received at least 1 dose of study medication.
Groups:
- Rocklatan (Latanoprost Mono): Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution, one drop in each eye in the evening for 12 weeks (Latanoprost Mono medical therapy regimen)
- Rocklatan (Latanoprost +1): Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution, one drop in each eye in the evening for 12 weeks (Latanoprost +1 medical therapy regimen)
- Rocklatan (Latanoprost +2): Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution, one drop in each eye in the evening for 12 weeks (Latanoprost +2 medical therapy regimen)
Period: Overall Study
Arm/Group | Rocklatan (Latanoprost Mono) | Rocklatan (Latanoprost +1) | Rocklatan (Latanoprost +2)
Started | 61 | 45 | 30
Completed | 54 | 37 | 25
Not Completed | 7 | 8 | 5
Not completed — Adverse Event | 4 | 4 | 0
Not completed — Patient Lost to Follow-Up | 0 | 0 | 1
Not completed — Patient Withdrawal | 2 | 4 | 2
Not completed — Investigator Decision | 1 | 0 | 1
Not completed — Enrolled in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All subjects who have received at least 1 dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocklatan (Latanoprost Mono) | Rocklatan (Latanoprost +1) | Rocklatan (Latanoprost +2) | Total
Number analyzed (Participants) | 61 | 45 | 30 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (11.2) | 71.1 (10.06) | 69.3 (11.60) | 69.0 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 23 | 14 | 69
  Male | 29 | 22 | 16 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 10 | 30
  Not Hispanic or Latino | 48 | 38 | 20 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 1 | 2 | 1 | 4
  Black or African American | 13 | 9 | 11 | 33
  White | 46 | 32 | 16 | 94
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Intraocular Pressure (IOP) at Week 12
Description: IOP was measured using Goldmann applanation tonometry at the Baseline and Week 12 visits. One eye (study eye) contributed data to this analysis. A negative value indicates an improvement in IOP. No hypothesis testing was prespecified for this endpoint.
Time Frame: Baseline (Day 0 pretreatment), Week 12
Population: All subjects that received at least 1 follow-up visit with a completed IOP measure and with complete data at both baseline and final visits.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Rocklatan Total: Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution, one drop in each eye in the evening for 12 weeks (Inclusive of all Latanoprost medical therapy regimens)
Arm/Group | Rocklatan (Latanoprost Mono) | Rocklatan (Latanoprost +1) | Rocklatan (Latanoprost +2) | Rocklatan Total
Number analyzed (Participants) | 54 | 37 | 25 | 116
percent change | -21.2 (17.46) | -15.7 (21.91) | -16.9 (17.31) | -18.5 (18.96)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of individual participation in the study, approximately 12 weeks (±7 days).
Description: An AE was defined as any untoward medical occurrence associated with the administration of the study intervention in humans, whether or not considered related to the study medication. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. This analysis population includes subjects who have received at least 1 dose of study medication.
Arm/Group | Rocklatan (Latanoprost Mono) | Rocklatan (Latanoprost +1) | Rocklatan (Latanoprost +2)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/45 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/45 | 1/30
Other Adverse Events (participants affected / at risk) | 9/61 | 10/45 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rocklatan (Latanoprost Mono) (N=61) | Rocklatan (Latanoprost +1) (N=45) | Rocklatan (Latanoprost +2) (N=30)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rocklatan (Latanoprost Mono) (N=61) | Rocklatan (Latanoprost +1) (N=45) | Rocklatan (Latanoprost +2) (N=30)
Conjunctival hyperaemia (Eye disorders) | 9 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT05283395/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT05283395/SAP_001.pdf